CLINICAL TRIAL: NCT05248230
Title: An Open-label, Phase 1/2 Trial of Gene Therapy 4D-710 in Adults With Cystic Fibrosis
Brief Title: 4D-710 in Adult Patients With Cystic Fibrosis
Acronym: CF
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: 4D Molecular Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 4D-710-C001
Record Dates: First submitted 2022-02-10; First posted 2022-02-21 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis Lung
Keywords: CF; Cystic Fibrosis; Gene Therapy
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 4D-710 Phase 1: Dose Exploration (Experimental): Participants who are ineligible for or intolerant of modulator therapy will receive one of various dose levels of 4D-710 to identify recommended phase 2 dose(s) for further evaluation.
  Interventions: Biological: 4D-710
- 4D-710 Phase 2: Dose Expansion (Experimental): Participants will receive a single inhalational administration of 4D-710 at the dose level(s) selected for dose expansion.
  Interventions: Biological: 4D-710
- 4D-710 Dose Exploration (Sub-Study) (Experimental): Participants who are on currently available CFTR modulator therapy will receive a dose of 4D-710 at various dose levels.
  Interventions: Biological: 4D-710

INTERVENTIONS:
Biological: 4D-710 — 4D-710 is an adeno-associated virus (AAV) gene therapy comprised of an AAV capsid variant (4D-A101) carrying a transgene cassette encoding human cystic fibrosis transmembrane conductance regulator with a deletion in the regulatory domain (CFTRΔR).

SUMMARY:
This is a Phase 1/2 multicenter, open-label, single dose trial of 4D-710 investigational gene therapy in adults with cystic fibrosis.

DETAILED DESCRIPTION:
This Phase 1/2 trial will evaluate the safety, tolerability, and preliminary efficacy of 4D-710, an investigational gene therapy, in adults with cystic fibrosis (CF) advanced lung disease who are ineligible or unable to tolerate CFTR modulator therapy. A sub-study will evaluate 4D-710 in a cohort of adults with CF advanced lung disease and/or frequent pulmonary exacerbation (PE) while on currently available CFTR modulator therapy.

ELIGIBILITY:
Key Inclusion Criteria (Primary Study):

1. 18 years and older
2. Confirmed diagnosis of cystic fibrosis (CF) and CF lung disease including:

   1. Sweat chloride ≥ 60 mmol/L
   2. Mutation Status

      * Bi-allelic mutations in the CFTR gene, or
      * Single mutation in the CFTR gene and clinical manifestations of CF lung disease
   3. Ineligible for CFTR modulator therapy, or previously received modulator therapy but discontinued due to adverse effects.
3. Forced expiratory volume in 1 second (FEV1) ≥ 50% and ≤ 90% of predicted (per Global Lung Function Initiative) at Screening
4. Resting oxygen saturation ≥ 92% on room air at Screening

Key Inclusion Criteria (Sub-Study):

1. 18 years and older
2. Confirmed diagnosis of cystic fibrosis (CF) and CF lung disease including:

   1. Sweat chloride ≥ 60 mmol/L
   2. Mutation Status

      * Bi-allelic mutations in the CFTR gene, or
      * Single mutation in the CFTR gene and clinical manifestations of CF lung disease
3. Currently on a stable dose of CFTR modulator therapy (elexacaftor/tezacaftor/ivacaftor) for a minimum of 60 days prior to Screening and agree to maintain current regimen through the 12-month Observation Period
4. FEV1 ≥ 40% and < 70% predicted (per Global Lung Function Initiative) at Screening, AND/OR experienced at least 2 pulmonary exacerbations in the last year requiring intravenous antibiotics

Key Exclusion Criteria (Primary and Sub Study):

1. Any prior gene therapy for any indication (Exception: mRNA-based therapies are not exclusionary)
2. Active Mycobacterium abscessus infection requiring ongoing treatment at Screening
3. Active allergic bronchopulmonary aspergillosis requiring management with systemic corticosteroids or antifungal therapy
4. Contraindication to systemic corticosteroid therapy
5. Requires chronic use of systemic corticosteroids or immunosuppressants to treat another condition
6. If no known diagnosis of cystic fibrosis related diabetes (CFRD), Type I, or Type II diabetes: Hemoglobin A1C ≥ 6.5% at Screening
7. If known diagnosis of CFRD, Type I or Type II diabetes: Hemoglobin A1C > 7.5% at Screening
8. Recent history of symptomatic hyperglycemia or unstable blood glucose levels as per Investigator's assessment
9. Other conditions that, in the Investigator's opinion, may interfere with management of corticosteroid-related hyperglycemia
10. Body Mass Index (BMI) < 16
11. Laboratory abnormalities at screening:

    * ALT, AST or GGT ≥ 3 × the upper limit of normal (ULN)
    * Total bilirubin ≥ 2 × ULN
    * Hemoglobin < 10 g/dL
12. Requirement for continuous or night-time oxygen supplementation
13. Known CF liver disease with evidence of multilobular cirrhosis
14. History of thrombosis (excluding catheter-related thrombosis) or conditions associated with increased risk of thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | 60 Months
  Safety and tolerability of 4D-710 following a single inhalation dose, as assessed by incidence and severity of treatment emergent adverse events, serious adverse events, and dose limiting toxicities, including clinically significant changes from baseline to scheduled time points in safety parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Zachary M Sellers, MD, PhD, Study Director — 4D Molecular Therapeutics
Locations (19):
- United States (19):
  - University of Alabama Child Health Research Unit, Birmingham, Alabama
  - The University of Arizona, Tucson, Arizona
  - University of California San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Miami Hospital, Miami, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Rainbow Babies and Children's Hospital/University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Penn State Health, Hershey, Pennsylvania
  - The Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Virginia Commonwealth University Health System, Richmond, Virginia
  - University of Washington Medical Center, Seattle, Washington

REFERENCES:
- [Derived] Calton MA, Croze RH, Sullivan TH, Collins SA, Tucker S, Whittlesey KJ, Kim DH, Nye JA, Beliakoff G, Quezada M, Burns C, Schmitt C, Klein A, Jia V, Kovacs L, Lauko D, Yoh K, Nguyen K, Barglow K, Gonzales J, Khoday D, Mason T, Delaria K, Bashour K, Kotterman M, Schaffer D, Song A, Francis P, Taylor-Cousar JL, Kirn D. Design and Characterization of 4D-710, an Aerosolized Gene Therapy for Cystic Fibrosis Lung Disease. Am J Respir Cell Mol Biol. 2025 Oct 22. doi: 10.1165/rcmb.2025-0243MA. Online ahead of print. PMID 41124321